CLINICAL TRIAL: NCT03627013
Title: A Prospective, Randomized, Single Blind, Multicentre Phase III Study on Organ Preservation With Custodiol-N Solution Compared With Custodiol Solution in Or-gan Transplantation (Kidney, Liver and Pancreas)
Brief Title: Custodiol-N Solution Compared With Custodiol Solution in Organ Transplantation (Kidney, Liver and Pancreas)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-N-KLP-TX-III/07-AT/17; 2017-002198-20 (EudraCT Number)
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Kidney Failure; Liver Failure, Chronic; Kidney-Pancreas Failure
MeSH Terms: conditions — Renal Insufficiency; End Stage Liver Disease | interventions — Custodiol-N solution; Bretschneider cardioplegic solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Kidney Custodiol-N (Experimental)
  Interventions: Drug: Custodiol-N Solution
- Kidney Custodiol (Active Comparator)
  Interventions: Drug: Custodiol HTK Solution
- Liver Custodiol-N (Experimental)
  Interventions: Drug: Custodiol-N Solution
- Liver Custodiol (Active Comparator)
  Interventions: Drug: Custodiol HTK Solution
- Kidney/Pancreas Custodiol-N (Experimental)
  Interventions: Drug: Custodiol-N Solution
- Kidney/Pancreas Custodiol (Active Comparator)
  Interventions: Drug: Custodiol HTK Solution

INTERVENTIONS:
Drug: Custodiol-N Solution — Perfusion
  Arms: Kidney Custodiol-N; Kidney/Pancreas Custodiol-N; Liver Custodiol-N
Drug: Custodiol HTK Solution — Perfusion
  Arms: Kidney Custodiol; Kidney/Pancreas Custodiol; Liver Custodiol

SUMMARY:
Synopsis Title of Study A prospective, randomized, single blind multicentre phase III study on organ preservation with Custodiol-N compared with Custodiol solution in organ transplantation (kidney, liver and pancreas)

Protocol number: CL-N-KLP-TX-III/07-AT/17

Trial design The study design is a prospective, randomized, single blind, multicentre, phase III comparison study of organ perfusion intended to demonstrate non-inferiority of Custodiol-N against Custodiol in organ transplantation of kidney, combined kidney-pancreas and liver.

Intended duration of study The overall duration for the trial is expected to be approximately 30 months. The du-ration of the trial for each subject is expected to be 3 months (transplantation and a follow-up period of 90 days).

Purpose of the study

The objective of this investigation is to demonstrate non-inferiority of graft preservation with Custodiol-N compared to Custodiol with respect to both graft function and injury after transplantation of kidney, liver or combined kidney-pancreas.

Patient selection The study population will be selected from patients who will undergo kidney, liver or combined kidney-pancreas transplantation. Patients of each gender will be included in the study.

Planned number of patients (recipients)

In total N=362 including:

Kidney 242 (including approx. 30 combined kidney-pancreas)

Liver 120

ELIGIBILITY:
Inclusion Criteria:

* All organs (kidney, combined kidney - pancreas and liver) Donor criteria

For All patients undergoing deceased donation:

- deceased adult (≥18 years) donors fulfilling the criteria for organ donation

For All patients undergoing living kidney donation:

- adult (≥18 years) living kidney donors fulfilling the criteria for organ donation

Patient (recipient) criteria

* recipients awaiting their transplant
* recipients ≥18 years
* recipients' signed informed consent before the transplantation Kidney / combined kidney - pancreas recipients
* n/a Liver recipient
* full organ transplantation

Exclusion Criteria:

* All organs (kidney, combined kidney - pancreas and liver) Donor criteria (not applicable for living kidney donors)
* - donors whose organs are all allocated out of retrieving study center
* general refusal of organ donation
* donation after cardiac death (DCD) Patient (recipient) criteria
* pregnant or lactating patients
* recipients participating in any interventional study (e.g. another study involving compound/interventions aimed at the reduction of preservation and / or ischemia / reperfusion injury)
* all combined allocations other than pancreas and kidney

Kidney / combined kidney -pancreas recipient

* double kidney transplantation
* pancreas retransplantation
* machine perfusion According to the KDIGO-Guidelines (2009) all patients with PRA >0% are only included in the living donation setting.

Liver recipient

* retransplantation
* machine perfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Kidney: - delayed graft function: Dialysis requirement during the first week af-ter transplantation | 7 days
Liver: - area under the curve (AUC) GPT (ALT) after transplantation during 7 days (minimum 1 measurement per day) | 7 days

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (4):
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Ordensklinikum Linz, Linz
  - Medical University Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No